CLINICAL TRIAL: NCT02779283
Title: A Phase Ib Feasibility Study of Personalized Kinase Inhibitor Therapy Combined With Induction in Acute Leukemias Who Exhibit In Vitro Kinase Inhibitor Sensitivity
Brief Title: Personalized Kinase Inhibitor Therapy Combined With Chemotherapy in Treating Patients With Newly Diagnosed Acute Myeloid Leukemia and Acute Lymphoblastic Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Stephen Spurgeon, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB00011766; NCI-2016-00083 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); IRB00011766 (Other: OHSU Knight Cancer Institute); P30CA069533 (NIH)
Record Dates: First submitted 2016-05-18; First posted 2016-05-20 (Estimated); Last update posted 2020-05-26 (Actual); Status verified 2020-02

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute | interventions — Cyclophosphamide; Cytarabine; Dasatinib; Dexamethasone; Calcium Dobesilate; auricularum; dexamethasone acetate; dexamethasone 21-phosphate; Doxorubicin; Idarubicin; idelalisib; Leucovorin; Methotrexate; merphos; Methylprednisolone Hemisuccinate; Methylprednisolone; ponatinib; Rituximab; CT-P10; ruxolitinib; Sorafenib; Sunitinib; Vincristine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Arm I (AML) (Experimental): Patients receive cytarabine IV continuously over 24 hours on days 1-7, and idarubicin IV over 30 minutes on days 1-3.Patients receive cyclophosphamide IV over 3 hours twice daily (BID) on days 1-3, vincristine sulfate IV on days 4 and 11, doxorubicin hydrochloride IV on day 4, dexamethasone PO on days 1-4 and 11-14, and rituximab IV on day 1 and 11 (day 11 only of course 1). Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Based on the results of the kinase inhibitor assay (In Vitro Kinase Inhibitor Assay), patients receive either sorafenib tosylate PO BID, sunitinib malate PO daily, dasatinib PO daily, ponatinib hydrochloride PO daily, ruxolitinib phosphate or idelalisib PO BID on days 8-28 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cytarabine; Drug: Dasatinib; Drug: Idarubicin; Drug: Idelalisib; Device: In Vitro Kinase Inhibitor Assay; Drug: Ponatinib Hydrochloride; Drug: Ruxolitinib Phosphate; Drug: Sorafenib Tosylate; Drug: Sunitinib Malate
- Arm II (ALL) (Experimental): Patients receive cytarabine IV over 2 hours BID on days 2-3, methotrexate IV over 2-22 hours on day 1, methylprednisolone sodium succinate IV BID on days 1-3, leucovorin calcium IV every 6 hours until methotrexate level is < 0.05 uM and rituximab IV on days 1 and 8. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity. Based on the results of the kinase inhibitor assay (In Vitro Kinase Inhibitor Assay), patients receive either sorafenib tosylate PO BID, sunitinib malate PO daily, dasatinib PO daily, ponatinib hydrochloride PO daily, ruxolitinib phosphate or idelalisib PO BID on days 8-28 in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Drug: Cytarabine; Drug: Dasatinib; Drug: Dexamethasone; Drug: Doxorubicin Hydrochloride; Drug: Idelalisib; Device: In Vitro Kinase Inhibitor Assay; Drug: Leucovorin Calcium; Drug: Methotrexate; Drug: Methylprednisolone Sodium Succinate; Drug: Ponatinib Hydrochloride; Biological: Rituximab; Drug: Ruxolitinib Phosphate; Drug: Sorafenib Tosylate; Drug: Sunitinib Malate; Drug: Vincristine Sulfate

INTERVENTIONS:
Drug: Cyclophosphamide — Given IV
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
  Arms: Arm II (ALL)
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Dasatinib — Given PO
  Other Names: BMS-354825; Sprycel
Drug: Dexamethasone — Given PO
  Other Names: Aacidexam; Adexone; Aknichthol Dexa; Alba-Dex; Alin; Alin Depot; Alin Oftalmico; Amplidermis; Anemul mono; Auricularum; Auxiloson; Baycuten; Baycuten N; Cortidexason; Cortisumman; Decacort; Decadrol; Decadron; Decalix; Decameth; Decasone R.p.; Dectancyl; Dekacort; Deltafluorene; Deronil; Desamethasone; Desameton; Dexa-Mamallet; Dexa-Rhinosan; Dexa-Scheroson; Dexa-sine; Dexacortal; Dexacortin; Dexafarma; Dexafluorene; Dexalocal; Dexamecortin; Dexameth; Dexamethasonum; Dexamonozon; Dexapos; Dexinoral; Dexone; Dinormon; Fluorodelta; Fortecortin; Gammacorten; Hexadecadrol; Hexadrol; Lokalison-F; Loverine; Methylfluorprednisolone; Millicorten; Mymethasone; Orgadrone; Spersadex; Visumetazone
  Arms: Arm II (ALL)
Drug: Doxorubicin Hydrochloride — Given IV
  Other Names: 5,12-Naphthacenedione, 10-[(3-amino-2,3,6-trideoxy-alpha-L-lyxo-hexopyranosyl)oxy]-7,8, 9,10-tetrahydro-6,8,11-trihydroxy-8-(hydroxyacetyl)-1-methoxy-, hydrochloride, (8S-cis)- (9CI); ADM; Adriacin; Adriamycin; Adriamycin Hydrochloride; Adriamycin PFS; Adriamycin RDF; ADRIAMYCIN, HYDROCHLORIDE; Adriamycine; Adriblastina; Adriblastine; Adrimedac; Chloridrato de Doxorrubicina; DOX; DOXO-CELL; Doxolem; Doxorubicin.HCl; Doxorubin; Farmiblastina; FI 106; FI-106; hydroxydaunorubicin; Rubex
  Arms: Arm II (ALL)
Drug: Idarubicin — Given IV
  Other Names: 4-Demethoxydaunomycin; 4-demethoxydaunorubicin; 4-DMDR
  Arms: Arm I (AML)
Drug: Idelalisib — Given PO
  Other Names: CAL-101; GS 1101; GS-1101; Phosphoinositide-3 Kinase Delta Inhibitor CAL-101; Zydelig
Device: In Vitro Kinase Inhibitor Assay — Correlative studies
  Other Names: Laboratory Biomarker Analysis
Drug: Leucovorin Calcium — Given IV
  Other Names: Adinepar; Calcifolin; Calcium (6S)-Folinate; Calcium Folinate; Calcium Leucovorin; Calfolex; Calinat; Cehafolin; Citofolin; Citrec; citrovorum factor; Cromatonbic Folinico; Dalisol; Disintox; Divical; Ecofol; Emovis; Factor, Citrovorum; Flynoken A; Folaren; Folaxin; FOLI-cell; Foliben; Folidan; Folidar; Folinac; Folinate Calcium; folinic acid; Folinic Acid Calcium Salt Pentahydrate; Folinoral; Folinvit; Foliplus; Folix; Imo; Lederfolat; Lederfolin; Leucosar; leucovorin; Rescufolin; Rescuvolin; Tonofolin; Wellcovorin
  Arms: Arm II (ALL)
Drug: Methotrexate — Given IV
  Other Names: Abitrexate; Alpha-Methopterin; Amethopterin; Brimexate; CL 14377; CL-14377; Emtexate; Emthexat; Emthexate; Farmitrexat; Fauldexato; Folex; Folex PFS; Lantarel; Ledertrexate; Lumexon; Maxtrex; Medsatrexate; Metex; Methoblastin; Methotrexate LPF; Methotrexate Methylaminopterin; Methotrexatum; Metotrexato; Metrotex; Mexate; Mexate-AQ; MTX; Novatrex; Rheumatrex; Texate; Tremetex; Trexeron; Trixilem; WR-19039
  Arms: Arm II (ALL)
Drug: Methylprednisolone Sodium Succinate — Given IV
  Other Names: A-MethaPred; Asmacortone; Cryosolona; Medrate; Metypred; Prednilem; Solu Moderin; Solu-Medrol; Solu-Medrone
  Arms: Arm II (ALL)
Drug: Ponatinib Hydrochloride — Given PO
  Other Names: AP24534 HCl; Iclusig
Biological: Rituximab — Given IV
  Other Names: ABP 798; BI 695500; C2B8 Monoclonal Antibody; Chimeric Anti-CD20 Antibody; CT-P10; IDEC-102; IDEC-C2B8; IDEC-C2B8 Monoclonal Antibody; MabThera; Monoclonal Antibody IDEC-C2B8; PF-05280586; Rituxan; Rituximab Biosimilar ABP 798; Rituximab Biosimilar BI 695500; Rituximab Biosimilar CT-P10; Rituximab Biosimilar GB241; Rituximab Biosimilar IBI301; Rituximab Biosimilar PF-05280586; Rituximab Biosimilar RTXM83; Rituximab Biosimilar SAIT101; RTXM83
  Arms: Arm II (ALL)
Drug: Ruxolitinib Phosphate — Given PO
  Other Names: INCB-18424 Phosphate; Jakafi
Drug: Sorafenib Tosylate — Given PO
  Other Names: BAY 43-9006 Tosylate; BAY 54-9085; Nexavar; sorafenib
Drug: Sunitinib Malate — Given PO
  Other Names: SU011248; SU11248; sunitinib; Sutent
Drug: Vincristine Sulfate — Given IV
  Other Names: Kyocristine; Leurocristine sulfate; Leurocristine, sulfate; Oncovin; Vincasar; Vincosid; Vincrex; Vincristine, sulfate
  Arms: Arm II (ALL)

SUMMARY:
This phase IB trial studies the feasibility of using a functional laboratory based study to determine how well the test can be used to select personalized kinase inhibitor therapy in combination with standard chemotherapy in treating patients with newly diagnosed acute myeloid leukemia (AML) and acute lymphoblastic leukemia (ALL). It also evaluates safety and potential efficacy. Kinase inhibitor is a type of substance that blocks an enzyme called a kinase. Human cells have many different kinase enzymes, and they help control important cell functions. Certain kinases are more active in some types of cancer cells and blocking them may help keep the cancer cells from growing. Testing samples of blood from patients with AML and ALL in the laboratory with kinase inhibitors may help determine which kinase inhibitor has more activity against cancer cells and which one should be combined with standard of care chemotherapy. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving a personalized kinase inhibitor therapy combined with standard chemotherapy may be a better treatment for AML and ALL.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine feasibility of using an in vitro small molecule inhibitor screen to select kinase inhibitors to add to standard chemotherapy induction in AML or ALL.

SECONDARY OBJECTIVES:

I. Determine the safety and tolerability of the addition of the kinase inhibitors when added to standard chemotherapy induction.

II. Evaluate overall objective response rates at completion of induction therapy.

III. Evaluate need for re-induction at day 14 (+/- 3 days) for AML. IV. Evaluate sensitivity to kinase inhibitors using our in vitro small molecule inhibitor screen in newly diagnosed AML/ALL.

V. Determine twelve-month overall survival.

TERTIARY OBJECTIVES:

I. Perform next-generation mutational analysis in primary leukemia samples from study subjects at baseline to establish a panel of known mutations for each subject and at the time of bone marrow recovery after induction chemotherapy to measure residual disease and evaluate utility of next-generation sequencing as a method compared to flow cytometry for minimal residual disease (MRD).

II. Evaluate pharmacokinetics for each individual kinase inhibitor. III. Determine if there is a cytogenetic or other risk group that has a higher rate of treatment failure or inability to obtain results from the small molecule inhibitor screen.

OUTLINE: Patients are assigned to 1 of 2 arms.

ARM I (AML): Patients receive cytarabine intravenously (IV) continuously over 24 hours on days 1-7, and idarubicin IV over 30 minutes on days 1-3.

ARM II (ALL) CYCLE A: Patients receive cyclophosphamide IV over 3 hours twice daily (BID) on days 1-3, vincristine sulfate IV on days 4 and 11, doxorubicin hydrochloride IV on day 4, dexamethasone PO on days 1-4 and 11-14, and rituximab IV on day 1 and 11 (day 11 only of course 1). Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

ARM II (ALL) CYCLE B: Patients receive cytarabine IV over 2 hours BID on days 2-3, methotrexate IV over 2-22 hours on day 1, methylprednisolone sodium succinate IV BID on days 1-3, leucovorin calcium IV every 6 hours until methotrexate level is < 0.05 uM and rituximab IV on days 1 and 8. Treatment repeats every 28 days for up to 4 courses in the absence of disease progression or unacceptable toxicity.

In all arms, based on the results of the kinase inhibitor assay, patients receive either sorafenib tosylate PO BID, sunitinib malate PO daily, dasatinib PO daily, ponatinib hydrochloride PO daily, ruxolitinib phosphate or idelalisib PO BID on days 8-28 in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 4-6 weeks, and then for a minimum of 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed AML or ALL, excluding acute promyelocytic leukemia (APL); for histological confirmation, a bone marrow biopsy and aspirate must be reviewed at Oregon Health & Science University (OHSU)
* Patients must have newly diagnosed AML or ALL without previous treatment; hydroxyurea will be allowed to control peripheral blast count as clinically indicated but would need to be stopped prior to initiation of tyrosine kinase inhibitor [TKI]); all-trans retinoic acid (ATRA) is permitted during the period prior to ruling out a diagnosis of APL; previous radiation treatment is allowable; patients must be deemed eligible for treatment with cytotoxic induction chemotherapy with cytarabine and idarubicin for AML or hyper-cyclophosphamide, dexamethasone, doxorubicin, vincristine sulfate (CVAD) for ALL; patients newly diagnosed with ALL must have received no prior treatment for their ALL with the exception of steroids (i.e. prednisone, dexamethasone); intrathecal methotrexate or cytarabine, allowed prior to and throughout the enrollment period for AML and ALL
* Subjects must be aged between >= 18 years and =< 64 for AML and > 40 and =< 64 for ALL
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* Total bilirubin < 2.0 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional ULN and thought to be due to hepatocellular dysfunction
* Potassium > lower limit of normal (LLN) or correctable with supplements prior to first dose of study medication
* Magnesium > LLN or correctable with supplements prior to first dose of study medication
* Total calcium (corrected for serum albumin) >= LLN or correctable with supplements prior to first dose of study medication
* Serum amylase and lipase =< 1.5 x institutional ULN
* International normalized ratio (INR) =< 2.0 or correctable to 2.0 with vitamin K therapy
* Corrected QT (QTc) =< 450 msec. for men or QTc =< 470 msec. for women
* Creatinine < 2.0 x ULN
* No clinically significant uncontrolled infections as determined by investigator
* Patients must be able to take oral medications
* Persons of reproductive potential must agree to an adequate method of contraception throughout treatment and for at least 4 weeks after study drug is stopped

  * Women of childbearing potential must have a negative serum or urine pregnancy test within 8 days prior to start of study drug administration
* Patients must be willing to accept blood product transfusions
* Ability to understand and the willingness to sign a written informed consent document and Health Insurance Portability and Accountability Act (HIPAA) documentation
* DRUG-SPECIFIC INCLUSION CRITERIA
* DASATINIB

  * Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 24 hours prior to the start of study drug
  * Women must not be breastfeeding
  * WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug, plus 30 days (duration of ovulatory cycle) for a total of 30 days post-treatment completion
  * Men who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug plus 90 days (duration of sperm turnover) for a total of 90 days post-treatment completion
  * Azoospermic males and WOCBP, who are not heterosexually active, are exempt from contraceptive requirements; however, WOCBP must still undergo pregnancy testing
  * Investigators shall counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and the implications of unexpected pregnancy; investigators shall advise WOCBP and male subjects who are sexually active with WOCBP on the use of highly effective contraception; highly effective methods of contraception have a failure rate of < 1% when used consistently and correctly
  * At a minimum, subjects must agree to the use of two methods of contraception, with one method being highly effective and the other method being either highly effective or less effective

Exclusion Criteria:

* Newly diagnosed AML patients who are identified with FLT3-ITD or tyrosine kinase domain (TKD) point mutation in the codon for an aspartate (D835) or an isoleucine (I836) residue
* Patients with a diagnosis of Philadelphia chromosome (Ph)+ ALL are not eligible
* Subjects who are currently receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to study agent or other agents used in the study
* Drugs that affect the cytochrome P450 family 3, subfamily A, polypeptide 4 (CYP3A4) systems are allowed but should be used with caution depending on specific kinase inhibitor used
* All outside study medications and supplements will be reviewed and monitored by the inpatient pharmacy team; patients will be discouraged from taking herbals and additional supplements
* Patients should not be prescribed concomitant medications that may contribute to prolonged QTc without consultation with the chemotherapy pharmacist; additional ECGs should be done at the investigator?s discretion to ensure the subject?s safety; drugs that are generally accepted to increase the risk of Torsades de Pointes, include (but not limited to):

  * Quinidine, procainamide, disopyramide
  * Amiodarone, ibutilide, dofetilide, sotalol
  * Erythromycin, clarithromycin
  * Chlorpromazine, mesoridazine, thioridazine, pimozide
  * Cisapride, bepridil, droperidol, methadone, arsenic, chloroquine, domperidone, halofantrine, levomethadyl, pentamidine, sparfloxacin, lidoflazine
* Left ventricular ejection fraction < 50%
* Uncontrolled intercurrent illness including but not limited to, symptomatic New York Heart Association (NYHA) class III congestive heart failure, uncontrolled angina pectoris, myocardial infarction or stroke within 6 months prior to enrollment, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients with a known human immunodeficiency virus (HIV) diagnosis are excluded from the study
* History of hypersensitivity to any of the kinase inhibitors included in this study
* Pregnant or lactating women are excluded from the study
* Diagnosed congenital long QT syndrome
* Any history of significant bleeding disorder unrelated to cancer, including any congenital bleeding disorder or any acquired bleeding disorder within one year of start of study
* Any history of clinically significant ventricular arrhythmia (such as ventricular tachycardia, ventricular fibrillation or torsade de pointes)
* Patients must not have clinically significant malabsorption syndrome or history
* All patients must discontinue anti-platelet agents or anticoagulants 7 days prior to initiation of study drug
* All patients with unhealed wounds or fistulas should not be given vascular endothelial growth factor (VEGF) inhibiting TKIs
* DRUG-SPECIFIC EXCLUSION CRITERIA
* PONATINIB

  * Patients with cytogenetically ?favorable risk' AML (core-binding factor leukemias) will not be enrolled on the ponatinib arm; testing with cytogenetics and fluorescence in situ hybridization (FISH) can establish this subtype within 7 days of the diagnostic bone marrow biopsy
  * History of acute pancreatitis within 1 year of study or history of chronic pancreatitis
  * Uncontrolled hypertriglyceridemia (triglycerides > 450 mg/dL)
  * Any history of myocardial infarction, stroke, or revascularization

    * Any history of venous thromboembolism including deep venous thrombosis or pulmonary embolism with the exception of upper Extremity/Line associated deep vein thrombosis (DVTs) which are adequately treated (line removed and/or patient anti-coagulated)
  * Uncontrolled hypertension (diastolic blood pressure > 90 mm Hg; systolic > 140 mm Hg); patients with hypertension should be under treatment on study entry to effect blood pressure control
* DASATINIB

  * Any history of second or third degree heart block (may be eligible if the subject currently has a pacemaker)
  * Known pulmonary arterial hypertension
  * Patients may not have clinically significant pleural or pericardial effusion per provider discretion
* SORAFENIB

  * Major surgery, open biopsy, or significant traumatic injury within 30 days
  * Non-healing wound, ulcer, or bone fracture
  * Thrombotic or embolic venous or arterial events, such as cerebrovascular accident, including transient ischemic attacks, arterial thrombosis, deep vein thrombosis and pulmonary embolism within the past 6 months
  * Upper Extremity/Line associated DVTs which are adequately treated (line removed and/or patient anticoagulated) are eligible
  * Uncontrolled hypertension
  * Active bleeding during screening
  * Hypersensitivity to sorafenib
* Idelalisib

  * Ongoing drug-induced liver injury, chronic active hepatitis C (hepatitis C virus [HCV]), chronic active hepatitis B (hepatitis B virus [HBV]), alcoholic liver disease, non-alcoholic steatohepatitis, primary biliary cirrhosis, extrahepatic obstruction caused by cholelithiasis, cirrhosis of the liver, portal hypertension, or history of autoimmune hepatitis
  * Ongoing symptomatic pneumonitis
  * Ongoing inflammatory bowel disease or autoimmune colitis
  * Ongoing cytomegalovirus (CMV) infection, treatment, or prophylaxis within the past 28 days prior to the screening test for active CMV
  * History of serious allergic reaction including anaphylaxis and epidermal necrolysis
* Ruxolitinib

  * Chronic active hepatitis C (HCV)

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2016-01-13 (Actual); Primary Completion 2018-04-19 (Actual); Study Completion 2018-09-20 (Actual)

PRIMARY OUTCOMES:
Proportion of subjects who start a targeted drug | On day 8
  A proportion of subjects whose targeted drug is identified and who start the kinase-inhibitor drug on day 8 will be estimated among all screened subjects along with the 95% confidence interval using the feasibility analysis set.

SECONDARY OUTCOMES:
Incidence of any grade 3 or higher dose limiting toxicity graded (DLT) according to Common Terminology Criteria for Adverse Events version 4.0 | Up to 6 weeks post-treatment
  DLT events will be tabulated and summarized. The incidence of DLT and its 95% confidence interval will be provided for the entire safety analysis set as well as for each targeted drug separately.
Overall objective response rates defined as morphologic, cytogenetic and molecular complete response (CR) rates at the end of induction period | At 14 days post-induction treatment
  The proportion and its 95% confidence interval will be provided for morphologic CR rate, cytogenetic CR rate, and molecular CR rate at the end of induction period. The descriptive statistics (mean, standard deviation, median, minimum and maximum) will be provided for % blasts at day 14 (+/- 3 days) for acute myeloid leukemia or show signs of disease progression requiring alternative treatment (re-induction) during the 21 day targeted treatment period (days 8-28) for acute lymphoblastic leukemia. The proportion and its 95% confidence interval will be provided for the proportion of patients who show sensitivity to each of the study drugs (i.e., IC50 < 20% of median IC50).
Proportion of patients who show sensitivity to each of the study kinase inhibitors | Baseline
  Measured as half maximal inhibitory concentration (IC50) < 20% of median IC50.
Overall survival | From date of the first treatment assessed up to 1 year
  Kaplan-Meier method will be used to estimate overall survival.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Spurgeon, Principal Investigator — OHSU Knight Cancer Institute
Locations (1):
- OHSU Knight Cancer Institute, Portland, Oregon, United States